CLINICAL TRIAL: NCT01076270
Title: A Pilot Study of Combined Plerixafor + Filgrastim for Mobilization of Peripheral Blood Stem Cells From Normal Donors
Brief Title: Plerixafor and Filgrastim For Mobilization of Donor Peripheral Blood Stem Cells Before A Donor Peripheral Blood Stem Cell Transplant in Treating Patients With Hematologic Malignancies
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding withdrawal
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2385.00; NCI-2010-00252 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2010-02-24; First posted 2010-02-26 (Estimated); Results first posted 2017-03-31 (Actual); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Accelerated Phase Chronic Myelogenous Leukemia; Adult Acute Lymphoblastic Leukemia in Remission; Adult Acute Myeloid Leukemia in Remission; Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Atypical Chronic Myeloid Leukemia, BCR-ABL Negative; Blastic Phase Chronic Myelogenous Leukemia; Chronic Phase Chronic Myelogenous Leukemia; de Novo Myelodysplastic Syndromes; Extranodal Marginal Zone B-cell Lymphoma of Mucosa-associated Lymphoid Tissue; Myelodysplastic/Myeloproliferative Neoplasm, Unclassifiable; Nodal Marginal Zone B-cell Lymphoma; Noncontiguous Stage II Adult Burkitt Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Mixed Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Small Cleaved Cell Lymphoma; Noncontiguous Stage II Adult Immunoblastic Large Cell Lymphoma; Noncontiguous Stage II Adult Lymphoblastic Lymphoma; Noncontiguous Stage II Grade 1 Follicular Lymphoma; Noncontiguous Stage II Grade 2 Follicular Lymphoma; Noncontiguous Stage II Grade 3 Follicular Lymphoma; Noncontiguous Stage II Mantle Cell Lymphoma; Noncontiguous Stage II Marginal Zone Lymphoma; Noncontiguous Stage II Small Lymphocytic Lymphoma; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Lymphoblastic Leukemia; Recurrent Adult Acute Myeloid Leukemia; Recurrent Adult Burkitt Lymphoma; Recurrent Adult Diffuse Large Cell Lymphoma; Recurrent Adult Diffuse Mixed Cell Lymphoma; Recurrent Adult Diffuse Small Cleaved Cell Lymphoma; Recurrent Adult Hodgkin Lymphoma; Recurrent Adult Immunoblastic Large Cell Lymphoma; Recurrent Adult Lymphoblastic Lymphoma; Recurrent Cutaneous T-cell Non-Hodgkin Lymphoma; Recurrent Grade 1 Follicular Lymphoma; Recurrent Grade 2 Follicular Lymphoma; Recurrent Grade 3 Follicular Lymphoma; Recurrent Mantle Cell Lymphoma; Recurrent Marginal Zone Lymphoma; Recurrent Mycosis Fungoides/Sezary Syndrome; Recurrent Small Lymphocytic Lymphoma; Refractory Chronic Lymphocytic Leukemia; Refractory Hairy Cell Leukemia; Refractory Multiple Myeloma; Relapsing Chronic Myelogenous Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Splenic Marginal Zone Lymphoma; Stage I Multiple Myeloma; Stage II Multiple Myeloma; Stage III Adult Burkitt Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Mixed Cell Lymphoma; Stage III Adult Diffuse Small Cleaved Cell Lymphoma; Stage III Adult Hodgkin Lymphoma; Stage III Adult Immunoblastic Large Cell Lymphoma; Stage III Adult Lymphoblastic Lymphoma; Stage III Chronic Lymphocytic Leukemia; Stage III Grade 1 Follicular Lymphoma; Stage III Grade 2 Follicular Lymphoma; Stage III Grade 3 Follicular Lymphoma; Stage III Mantle Cell Lymphoma; Stage III Marginal Zone Lymphoma; Stage III Multiple Myeloma; Stage III Small Lymphocytic Lymphoma; Stage IV Adult Burkitt Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Mixed Cell Lymphoma; Stage IV Adult Diffuse Small Cleaved Cell Lymphoma; Stage IV Adult Hodgkin Lymphoma; Stage IV Adult Immunoblastic Large Cell Lymphoma; Stage IV Adult Lymphoblastic Lymphoma; Stage IV Chronic Lymphocytic Leukemia; Stage IV Grade 1 Follicular Lymphoma; Stage IV Grade 2 Follicular Lymphoma; Stage IV Grade 3 Follicular Lymphoma; Stage IV Mantle Cell Lymphoma; Stage IV Marginal Zone Lymphoma; Stage IV Small Lymphocytic Lymphoma
MeSH Terms: conditions — Leukemia, Myeloid, Accelerated Phase; Congenital Abnormalities; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Mycosis Fungoides; Sezary Syndrome; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Hairy Cell; Multiple Myeloma | interventions — plerixafor; Filgrastim; Granulocyte Colony-Stimulating Factor; Peripheral Blood Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Filgrastim and plerixafor for PBSC mobilization (Experimental): Donors receive filgrastim subcutaneously (SC) and plerixafor SC on day -14 and undergo leukapheresis to collect peripheral blood stem cells (PBSC) on day -13. These cells are frozen to preserve them. Treatment modifications may apply according to sufficient collection of PBSC. Patients receive standard high-dose conditioning and undergo allogeneic PBSC transplantation on day 0 using the previously frozen cells.
  After completion of study treatment, donors are followed up 1 day after the last stem cell donation.
  Interventions: Drug: plerixafor; Biological: filgrastim; Procedure: peripheral blood stem cell transplantation; Procedure: allogeneic hematopoietic stem cell transplantation

INTERVENTIONS:
Drug: plerixafor — Given SC
  Other Names: AMD 3100; Mozobil
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen
Procedure: peripheral blood stem cell transplantation — Infusion of peripheral blood stem cells
  Other Names: PBPC transplantation; PBSC transplantation; peripheral blood progenitor cell transplantation; transplantation, peripheral blood stem cell
Procedure: allogeneic hematopoietic stem cell transplantation — Infusion of hematopoietic stem cells

SUMMARY:
RATIONALE: Giving chemotherapy and total-body irradiation (TBI) before a donor peripheral blood stem cell transplant helps stop the growth of cancer cells and helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they will help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Giving colony-stimulating factors, such as filgrastim (G-CSF) and plerixafor, to the donor helps the stem cells move (mobilization) from the bone marrow to the blood so they can be collected and stored.

PURPOSE: This clinical trial is studying giving plerixafor and filgrastim together for mobilization of donor peripheral blood stem cells before a peripheral blood stem cell transplant in treating patients with hematologic malignancies

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. The percentage of normal donors who collect at least 2 x 10^6 CD34 cells/kg recipient weight on day 1 after administration of combined filgrastim and plerixafor.

SECONDARY OBJECTIVES:

I. Measuring CD34+ cells/ul in peripheral blood of donors 11, 15, 24 and 36 hours post dosing.

II. Tolerance and safety of combined filgrastim and Plerixafor in normal donors.

III. Engraftment of filgrastim/plerixafor mobilized stem cells in allogeneic recipients.

IV. Acute and chronic graft-versus-host disease (GVHD) following the use of filgrastim/plerixafor mobilized stem cells.

V. Yield of CD34+ cells based on donor weight.

OUTLINE: Donors receive filgrastim subcutaneously (SC) and plerixafor SC on day -14 and undergo leukapheresis to collect peripheral blood stem cells (PBSC) on day -13. These cells are frozen to preserve them. Treatment modifications may apply according to sufficient collection of PBSC. Patients receive standard high-dose conditioning and undergo allogeneic PBSC transplantation on day 0 using the previously frozen cells.

After completion of study treatment, donors are followed up 1 day after the last stem cell donation.

ELIGIBILITY:
Inclusion Criteria:

* Hematologic malignancy considered eligible and suitable for allogeneic stem cell transplantation (syngeneic transplantation is acceptable); diagnoses include acute myeloid or lymphoid leukemias, chronic myeloid or lymphoid leukemias, multiple myeloma, lymphoma or myelodysplasia; subjects suitable for this study will primarily receive transplant on a standard treatment plan (non research regimen)
* Organ function, performance status and age suitable for an ablative regimen consisting of TBI >= 10Gy or a chemotherapy regimen consisting of busulphan and cyclophosphamide (BuCY) or busulphan and melphalan (BuMel)
* Availability of a fully matched sibling donor
* Ability to understand and willingness to sign an informed consent
* No uncontrolled infections
* DONOR: Human leukocyte antigen (HLA) identical sibling donor
* DONOR: >= 18 years
* DONOR: No unacceptable risk to donor due to pre-existing illness
* DONOR: Must have suitable antecubital veins for leukapheresis venipuncture; donors who will require a temporary, Mahurkar-type catheter are not eligible
* DONOR: Ability and willingness to sign an informed consent document

Exclusion Criteria:

* Eligible for and willingness to participate in any research study of transplant regimens
* Eligible for and willingness to participate in a non ablative transplant regimen
* Human immunodeficiency virus (HIV) seropositive
* Pregnancy
* DONOR: HIV seropositive
* DONOR: Contraindication or hypersensitivity to filgrastim or plerixafor
* DONOR: Hepatitis A, B, C seropositive
* DONOR: Pregnant or lactating females
* DONOR: Liver function studies > 2 times the upper limit of normal (ULN) at evaluation, Creatinine > 2, pulmonary function diffusing lung capacity for carbon monoxide (DLCO) < 50% (if specifically evaluated), cardiac ejection fraction < 50% (if specifically evaluated)
* DONOR: Any known ventricular arrhythmia

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-06; Primary Completion 2011-01 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Bensinger, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (1):
- Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Filgrastim and Plerixafor for PBSC Mobilization: Donors receive filgrastim subcutaneously (SC) and plerixafor SC on day -14 and undergo leukapheresis to collect peripheral blood stem cells (PBSC) on day -13. These cells are frozen to preserve them. Treatment modifications may apply according to sufficient collection of PBSC. Patients receive standard high-dose conditioning and undergo allogeneic PBSC transplantation on day 0 using the previously frozen cells.
  After completion of study treatment, donors are followed up 1 day after the last stem cell donation.
  plerixafor: Given SC
  filgrastim: Given SC
  peripheral blood stem cell transplantation: Infusion of peripheral blood stem cells
  allogeneic hematopoietic stem cell transplantation: Infusion of hematopoietic stem cells
Period: Overall Study
Arm/Group | Filgrastim and Plerixafor for PBSC Mobilization
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Filgrastim and Plerixafor for PBSC Mobilization
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Successful Collection of Stem Cells
Description: Percentage of donors from whom at least 2 x 10^6 CD34+ cells/kg body weight were collected based on actual recipient body weight
Time Frame: At the end of apheresis for cell collection
Population: Study terminated early. Results are for the one donor enrolled.
Measure: Count of Participants; unit: Participants
Arm/Group | Filgrastim and Plerixafor for PBSC Mobilization
Number analyzed (Participants) | 1
Participants | 1

2. Secondary Outcome: CD34-positive Cells Collected
Description: Number of CD34-positive cells collected per kg recipient body weight
Time Frame: At the end of apheresis for cell collection
Population: Trial terminated; only one patient enrolled
Measure: Number; unit: CD34-positive cells collected/kg
Arm/Group | Filgrastim and Plerixafor for PBSC Mobilization
Number analyzed (Participants) | 1
CD34-positive cells collected/kg | 4,760,000

ADVERSE EVENTS:
Time Frame: From the first dose of study drug to one week after the last clinic visit. The last clinic visit typically occurs the day after stem cell collection is completed.
Arm/Group | Filgrastim and Plerixafor for PBSC Mobilization
All-Cause Mortality (participants affected / at risk) | 1/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 1/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Filgrastim and Plerixafor for PBSC Mobilization (N=1)
Lightheadedness (General disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Only one patient was enrolled in this trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less